CLINICAL TRIAL: NCT01085123
Title: An Open Label, Positron Emission Tomography (PET) Study With [11C]AZ10419369 to Determine Central 5-HT1B Receptor Occupancy of ZOMIG® Rapimelt (Zolmitriptan) in Healthy Male Volunteers
Brief Title: Determine Central 5-HT1B Receptor Occupancy of ZOMIG® Rapimelt (Zolmitriptan) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1220C00005
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Migraine
Keywords: Migraine; ZOMIG® Rapimelt
MeSH Terms: conditions — Migraine Disorders | interventions — zolmitriptan; 5-methyl-8-(4-methyl-piperazin-1-yl)-4-oxo-4H-chromene-2-carboxylic acid (4-morpholin-4-yl-phenyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PET 1: baseline, PET 2: 10 mg Zomig® Rapimelt, PET 3: 5 mg ZOMIG® Rapimelt, PET 4 2.5 mg ZOMIG® Rapimelt
  Interventions: Drug: Rapimelt; Drug: [11C]AZ10419369

INTERVENTIONS:
Drug: Rapimelt — oral tablet , 2.5 and 5 mg, single dose. 10 mg (2x5 mg) visit 3, 5 mg visit 4, 2.5 mg visit 5.
  Other Names: ZOMIG®
Drug: [11C]AZ10419369 — solution for iv injection. Will be injected within 2 to 5 hours after administration of ZOMIG® Rapimelt

SUMMARY:
The purpose of this study is to determine the central 5-HT1B receptor occupancy of ZOMIG® Rapimelt (zolmitriptan) in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between ≥19 and ≤30 kg/m2.

Exclusion Criteria:

* A history or presence of neurological, haematological, psychiatric, gastrointestinal, hepatic, pulmonary, renal disease
* Use of drugs that induce the liver drug metabolising enzymes within 4 weeks before first PET

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine zolmitriptan and/or its active metabolite 183C91 occupancy at 5-HT1B receptors in the living human brain | The first PET measurement will serve as a baseline assessment. The second, third and fourth PET measurements will be performed after oral administration of ZOMIG® Rapimelt (10 mg, 5 mg and 2.5 mg, respectively).

SECONDARY OUTCOMES:
To describe the relation between Zomig® Rapimelt dose and 5-HT1B receptor occupancy | The second, third and fourth PET measurements will be performed after oral administration of ZOMIG® Rapimelt (10 mg, 5 mg and 2.5 mg, respectively). Imaging data analysis will be performed after each PET measurement
To describe the relation between plasma concentrations of zolmitriptan and 183C91 and 5-HT1B receptor occupancy | For each of 3 visits venous blood for zolmitriptan and 183C91 PK analyses taken before drug administration and at 3 time points during PET examination: start, middle and end, ie, at 0, +30 and + 63 minutes relative to injection of the radioli

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kanes, Study Director — AstraZeneca; Wolfgang Kühn, Principal Investigator — Quintiles AB Phase I Services; Brendan Smyth, Study Chair — AstraZeneca
Locations (1):
- Research Site, Uppsala, Sweden